CLINICAL TRIAL: NCT03299478
Title: Clinical Implementation of TNM-immunoscore in Resected Non-small Cell Lung Cancer
Acronym: TNM-I
Status: Active, not recruiting | Type: Observational
Sponsor: University Hospital of North Norway (Other)
Collaborators: Norwegian Cancer Society (Other); Northern Health Authority (Other Government); St. Olavs Hospital (Other); Rigshospitalet, Denmark (Other); Odense University Hospital (Other); Oslo University Hospital (Other); University of Tromso (Other)
Responsible Party: Sponsor
Other Study IDs: 2016/714
Record Dates: First submitted 2017-09-27; First posted 2017-10-03 (Actual); Last update posted 2024-06-11 (Actual); Status verified 2024-05

CONDITIONS: Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples With DNA — Tumor specimen Blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- NSCLC patients: Resected NSCLC patients with curative intent
  Interventions: Other: Will look for immune infiltration

INTERVENTIONS:
Other: Will look for immune infiltration

SUMMARY:
The purpose of this study is to validate TNM-Immunoscore in resected non-small cell lung cancer.

DETAILED DESCRIPTION:
The main aim is to validate the most promising T-cell marker candidates from earlier studies in a prospective multicenter study to establish a prognostic TNM-Immunoscore.

The investigators will include around 1000 stage I-IIIA patients from various centers in Scandinavia. The investigators will also collect demographic and clinicopathological data, blood and tissues in a database and biobank. Candidate T-cell markers will be analyzed by immunohistochemistry for validation and by other methods for exploration of their impact on prognosis

ELIGIBILITY:
Inclusion Criteria:

* resectable NSCLC
* Age 18 and above
* no other malignancy last 5 years
* informed consent

Exclusion Criteria:

* multiple tumor foci
* preoperative chemo- or radiotherapy
* non-NSCLC histology
* no tissue available for study
* metastasis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Pasients coming for resection of primary NSCLC with a curative intent
Sampling Method: Probability Sample
Enrollment: 865 (Actual)
Dates: Start 2016-11-28 (Actual); Primary Completion 2027-02-01 (Estimated); Study Completion 2027-02-01 (Estimated)

PRIMARY OUTCOMES:
Overall survival | 5 year follow-up
  Overall survival in the 1) overall population and in the 2) squamous cell carcinoma and 3) adenocarcinoma subgroups.

SECONDARY OUTCOMES:
TTR | 5 year follow-up
  Time to recurrence in the 1) overall population and in the 2) squamous cell carcinoma and 3) adenocarcinoma subgroups.
Disease-specific survival | 5 year follow-up
  Disease specific survival in the 1) overall population and in the 2) squamous cell carcinoma and 3) adenocarcinoma subgroups.

CONTACTS AND LOCATIONS:
Overall Officials: Lill-Tove R Busund, MD, PhD, Principal Investigator — University Hospital of North Norway; Sigve Andersen, MD,PhD, Principal Investigator — University Hospital of North Norway; Tom Dønnem, MD,PhD, Principal Investigator — University Hospital of North Norway
Locations (5):
- Denmark (2):
  - Rigshospitalet, Copenhagen, København Ø
  - Odense Universitetshospital, Odense
- Norway (3):
  - Oslo University Hospital, Oslo
  - University Hospital of North Norway, Tromsø
  - St.Olav Hospital, University Hospital of Trondheim, Trondheim

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Donnem T, Kilvaer TK, Andersen S, Richardsen E, Paulsen EE, Hald SM, Al-Saad S, Brustugun OT, Helland A, Lund-Iversen M, Solberg S, Gronberg BH, Wahl SG, Helgeland L, Flotten O, Pohl M, Al-Shibli K, Sandanger TM, Pezzella F, Busund LT, Bremnes RM. Strategies for clinical implementation of TNM-Immunoscore in resected nonsmall-cell lung cancer. Ann Oncol. 2016 Feb;27(2):225-32. doi: 10.1093/annonc/mdv560. Epub 2015 Nov 16. PMID 26578726
- [Result] Rakaee M, Andersen S, Giannikou K, Paulsen EE, Kilvaer TK, Busund LR, Berg T, Richardsen E, Lombardi AP, Adib E, Pedersen MI, Tafavvoghi M, Wahl SGF, Petersen RH, Bondgaard AL, Yde CW, Baudet C, Licht P, Lund-Iversen M, Gronberg BH, Fjellbirkeland L, Helland A, Pohl M, Kwiatkowski DJ, Donnem T. Machine learning-based immune phenotypes correlate with STK11/KEAP1 co-mutations and prognosis in resectable NSCLC: a sub-study of the TNM-I trial. Ann Oncol. 2023 Jul;34(7):578-588. doi: 10.1016/j.annonc.2023.04.005. Epub 2023 Apr 24. PMID 37100205